CLINICAL TRIAL: NCT00022685
Title: A Phase III Clinical Trial of Immunotherapy With Humanized LL2 IgG (Epratuzumab) in Patients With Low-Grade Follicular, B-Cell Non-Hodgkin's Lymphoma Refractory to Rituxan (Rituximab)
Brief Title: Epratuzumab in Treating Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068842; UCLA-0009041; IM-T-hLL2-07; UCLA-BB-IND-7124; NCI-G01-2004
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2003-04

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — epratuzumab

INTERVENTIONS:
Biological: epratuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies such as epratuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase III trial to determine the effectiveness of epratuzumab in treating patients who have low-grade non-Hodgkin's lymphoma that has not responded to chemotherapy or rituximab.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of epratuzumab in patients with rituximab-refractory low-grade follicular B-cell non-Hodgkin's lymphoma.
* Confirm the convenient administration of this drug in this patient population.
* Determine the efficacy of this drug in terms of objective response rate in these patients.
* Determine the duration of response and time to progression in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive epratuzumab IV over 15-60 minutes on days 1, 8, 15, and 22.

Patients are followed every 8 weeks for 10 months and then every 3 months for up to 4 years.

PROJECTED ACCRUAL: Approximately 30-100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade follicular B-cell non-Hodgkin's lymphoma

  * Small cleaved cell OR
  * Mixed cell
* The following are ineligible:

  * Primary CNS lymphoma
  * HIV lymphoma
  * Richter's lymphoma
  * Bulky disease (any single mass greater than 10 cm)
  * Pleural effusion with positive cytology for lymphoma
* Failed prior standard chemotherapy for non-Hodgkin's lymphoma
* Refractory to at least 1 prior treatment with rituximab

  * Disease progression or failure to achieve objective response within 6 months of beginning rituximab therapy
* At least 1 bidimensionally measurable lesion

  * At least 1.5 cm by CT scan NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%
* ECOG 0-2

Life expectancy:

* At least 4 months

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 50,000/mm^3
* Hemoglobin at least 8 g/dL
* Transfusion independent

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)*
* Alkaline phosphatase less than 2 times ULN*
* AST less than 2 times ULN* NOTE: *Unless lymphoma-related

Renal:

* Creatinine no greater than 1.5 times ULN unless lymphoma-related

Other:

* No other malignancy within the past 5 years except squamous or basal cell skin cancer or carcinoma in situ of the cervix
* No other serious condition or infection that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 12 weeks since prior autologous stem cell transplantation
* No prior radioimmunoconjugate therapies

Chemotherapy:

* See Disease Characteristics
* No more than 4 prior treatment regimens
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* At least 2 weeks since prior corticosteroids
* No concurrent steroids

Radiotherapy:

* See Biologic therapy
* At least 4 weeks since prior radiotherapy to target lesion

Surgery:

* At least 4 weeks since prior major surgery unless recovered

Other:

* At least 4 weeks since prior experimental therapies
* No other concurrent investigational or therapeutic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Rosen, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States